CLINICAL TRIAL: NCT00215371
Title: Study in Patients With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dey (Industry)
Responsible Party: Director, Clinical Affairs, Dey
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DL-050
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2010-11-11 (Estimated); Status verified 2008-02

CONDITIONS: Asthma
Keywords: Asthma; Pediatric; Formoterol Fumarate; Foradil
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol Fumarate

SUMMARY:
The purpose of this study is to determine which dose of the investigational drug is safest and most effective compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Require the regular use of an inhaled beta-2-selective adrenergic agent.
* No clinically significant abnormalities on the medical history, physical examination, and clinical laboratory tests.

Exclusion Criteria:

* Active acute or chronic disorders of the respiratory system within one month prior to screening.
* Smoking history within the past 12 months or greater than a lifetime 10 pack-year smoking history.
* Debilitating systemic and/or life-threatening diseases.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32
Dates: Start 2002-07; Primary Completion 2002-10 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Primary: The primary efficacy outcome is measure of lung function.

SECONDARY OUTCOMES:
Secondary: Change in lung function will be examined as a secondary efficacy outcome, as well as vital signs, physical examination, adverse event reporting,etc.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Long Beach, California
  - Research Site, Medford, Oregon